CLINICAL TRIAL: NCT02361034
Title: A Two-Part, Phase I Study of Orally Administered GRC 27864, a Novel, Microsomal Prostaglandin E Synthase-1 Enzyme (mPGES-1) Inhibitor, to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses in Healthy Subjects (Part 1), and of Multiple Doses in Elderly Subjects (Part 2)
Brief Title: To Evaluate Safety, Tolerability and Pharmacokinetics of GRC 27864 in Healthy Subjects and Elderly Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GRC 27864-102; 2014-001932-13 (EudraCT Number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Safety and pharmacokinetics of drug in healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GRC 27864 (Active Comparator): Test treatment GRC 27864
  Interventions: Drug: GRC 27864
- Placebo (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRC 27864
  Arms: GRC 27864
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multiple Ascending dose (MAD) study with GRC 27864 in Healthy and Elderly Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged ≥18 to <55 years (> 65 years for elderly cohort) at the time of informed consent
2. Body mass index (BMI) within the range 18.5-32 kg/m2 (inclusive); weight must be >50 kg
3. Subjects who are healthy and free from clinically significant illness or disease
4. Females must be of non-childbearing potential, surgically sterile.
5. Male subjects whose partners are of childbearing potential or have undergone tubal ligation must agree to use 2 highly effective methods of contraception

Exclusion Criteria:

1. Systolic blood pressure (SBP) <90 mmHg or >140 mmHg, diastolic blood pressure (DBP) <45 mmHg or >90 mmHg, resting pulse rate <40 beats per minute (bpm) or >100 bpm
2. Subjects who have the presence of active peptic ulcer disease, gastrointestinal (GI) bleeding, chronic gastritis, inflammatory bowel disease, chronic diarrhoea or positive 13C urea breath/faecal test for Helicobacter pylori at Screening.
3. Subjects with inherited or acquired disorders of platelet function, bleeding or coagulation.
4. Presence of any clinically relevant acute or chronic disease that could interfere with the subject's safety during the clinical study, expose the subject to undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of TEAEs and serious adverse events (SAEs) after multiple oral doses of GRC 27864 in healthy adult and elderly subjects | Baseline upto 42 days after administration of the study drug.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Time to Maximum Concentration (Tmax) of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Area Under Curve [AUC0-t and AUC0-tau] of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Half-life (t½) of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Volume of distribution (V)/bioavailability (F) of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Clearance (CL)/F of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Observed accumulation ratio (Rac) of GRC 27864 and its metabolite GRC 27884 following multiple doses in healthy adult subjects and elderly subjects. | Predose and postdose from 0.25 to 48 hrs and from Day 1 to day 28
Cerebrospinal fluid (CSF) concentrations of GRC 27864 and its metabolite GRC 27884 (CmaxCSF) following multiple doses to healthy adult subjects | 6 hours, and 24 hours postdose on Day 26

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, Principal Investigator — Medical Director
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, Yorkshire, United Kingdom